CLINICAL TRIAL: NCT00763698
Title: QuickFlex Micro Model 1258T Left Heart Pacing Lead
Brief Title: Safety and Efficacy Study of the QuickFlex Micro Model 1258T Left Heart Pacing Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD 435
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Results first posted 2011-11-04 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Left heart pacing lead; Cardiac resynchronization therapy (CRT); Heart failure; ICD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QuickFlex micro 1258T left heart lead (Experimental)
  Interventions: Device: QuickFlex Micro Model 1258T Left Heart Lead

INTERVENTIONS:
Device: QuickFlex Micro Model 1258T Left Heart Lead — Implantation of QuickFlex Micro 1258T left heart lead in combination with a CRT-D system.
  Other Names: Model 1258T left heart pacing lead

SUMMARY:
This is a prospective, multi-center non-randomized clinical study to evaluate the safety and efficacy of the QuickFlex Micro Model 1258T left ventricular lead in a heart failure patient population. The study will be conducted at a maximum of 20 investigational centers located in the United States and a total of 68 patients will be enrolled.

DETAILED DESCRIPTION:
The investigational left heart lead, QuickFlex Model 1258T, will be implanted with a legally marketed St. Jude Medical cardiac resynchronization therapy implantable cardioverter defibrillator (CRT-D) device.

Patients will be followed at Pre-Discharge, 1-Month, 3-Month,and then every 6 months until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Approved indication for CRT-D system

Exclusion Criteria:

* Previous cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 3 months of enrollment
* Previous left ventricular (LV) lead implant
* Have had a heart attack,unstable angina or cardiac revascularization (percutaneous transluminal coronary angioplasty (PTCA),coronary artery bypass grafting (CABG), Stent) within 40 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Shipman, Study Director — Abbott Medical Devices
Locations (13):
- United States (13):
  - University Hospital-University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Cardiology, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Glendale Memorial Hospital and Medical Center, Glendale, California
  - Regional Cardiology Associates, Sacramento, California
  - Midwest Heart Foundation, Lombard, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Thoracic Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - St. Francis Hospital, Roslyn, New York
  - EMH Regional Medical Center, Elyria, Ohio
  - St. Thomas Hospital, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 18 investigational centers located in the United States (US). The first patient was enrolled on October 30, 2008 and follow up was completed on May 31, 2009.
Pre-assignment Details: All patients were included in the study analysis with the exception of patients who underwent unsuccessful implantation of the 1258T lead system. These patients were followed for a period of 30 days and then were withdrawn from the study.
Groups:
- QuickFlex Micro 1258T Left Heart Lead: All patients received a QuickFlex Micro 1258T left heart lead and were evaluated for freedom from left ventricular lead complications at 3 months. Left ventricular lead related complications is defined as any adverse event related to the left ventricular lead that requires an invasive intervention.
Period: Overall Study
Arm/Group | QuickFlex Micro 1258T Left Heart Lead
Started | 86
Completed | 76
Not Completed | 10
Not completed — Unsuccessful Implant | 5
Not completed — Death | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | QuickFlex Micro 1258T Left Heart Lead
Number analyzed (Participants) | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 57
Region of Enrollment [Number; unit: participants]
  United States | 86

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Left Ventricular Lead-related Complications
Description: A Kaplan-Meier survival analysis was carried out for left ventricular lead related complications through 3 months. Percentage of patients who remained free from complications at 3 months was reported.
Time Frame: 3 months
Population: Analysis was conducted on the 81 patients with a successful left ventricular lead implant.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | QuickFlex Micro 1258T Left Heart Lead
Number analyzed (Participants) | 81
percent of participants | 100 [100 to 100]
Statistical Analysis 1: Comparison: QuickFlex Micro 1258T Left Heart Lead; The objective performance criteria established for freedom from left ventricular lead related complications at 3 months was greater than 80%. At least 80% of the patients were required to be free from left venticular lead related complications at 3 months; Test type: Superiority or Other; Kaplan-Meier Survival Analysis; Objective Performance Criteria = 80, 95% CI 1-sided [lower limit 5]

2. Primary Outcome: Percentage of Successful Left Ventricular Lead Implants
Description: Left ventricular lead implant success rate was calculated as the total number of patients who had a successful implant of the left ventricular QuickFlex Micro Model 1258T lead divided by the total number of patients who had an attempted implant. A successful implant was defined as the placement of the left ventricular lead in the coronary sinus for the purposes of pacing of the left ventricle with connection to the pulse generator.
Time Frame: 3 months
Population: All patients with an implant or attempted implant were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QuickFlex Micro 1258T Left Heart Lead
Number analyzed (Participants) | 86
percentage of participants | 94 [87 to 100]
Statistical Analysis 1: Comparison: QuickFlex Micro 1258T Left Heart Lead; Test type: Superiority or Other; Wilson score interval method; Objective Performance Criteria = 80, 97.5% CI 1-sided [lower limit 2.5]

3. Primary Outcome: Left Ventricular Bipolar Pacing Capture Threshold (Volts)
Description: The mean left ventricular capture threshold (amount of energy needed to pace the heart) is reported. An overall mean capture threshold of < 3 volts is required to meet this endpoint.
Time Frame: 3 months
Population: This effectiveness endpoint was carried out on the first 16 patients who had a LV lead bipolar pacing capture threshold measurement at 3 months at 0.5 ms pulse width. This patient cohort is referred to as the "Primary Pacing Capture Threshold Patient Cohort".
Measure: Mean (Standard Deviation); unit: volts
Groups:
- QuickFlex Micro 1258T Left Heart Leads: Patients included in this analysis include the first 16 patients to provide LV lead bipolar pacing capture threshold data at 3 months with a pulse width of 0.5 ms.
Arm/Group | QuickFlex Micro 1258T Left Heart Leads
Number analyzed (Participants) | 16
volts | 1.1 (0.3)

ADVERSE EVENTS:
Time Frame: Data was collected from the time the first patient was enrolled until follow up was completed; a total of 7 months.
Arm/Group | QuickFlex Micro 1258T Left Heart Lead
Serious Adverse Events (participants affected / at risk) | 4/86
Other Adverse Events (participants affected / at risk) | 20/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QuickFlex Micro 1258T Left Heart Lead (N=86)
Cardiac vein thrombus (Cardiac disorders) | 1 (1)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1)
Right ventricular lead dislodgement/migration (Surgical and medical procedures) | 1 (1)
Right ventricular lead cardiac perforation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QuickFlex Micro 1258T Left Heart Lead (N=86)
Cardiac vein thrombus (Cardiac disorders) | 1 (1)
Hematoma (Skin and subcutaneous tissue disorders) | 4 (4)
High defibrillation threshold (Cardiac disorders) | 3 (3)
Hypotension (Cardiac disorders) | 1 (1)
Left ventricular lead dislodgement/migration (Surgical and medical procedures) | 1 (1)
Elevated left ventricular pacing threshold (Cardiac disorders) | 1 (1)
Phrenic Nerve/Diaphragmatic Nerve stimulation (Surgical and medical procedures) | 10 (10)
Right atrial lead undersensing (Cardiac disorders) | 1 (1)
Device pocket stimulation (Surgical and medical procedures) | 1 (1)
Therapy for non-ventricular rhythm (Cardiac disorders) | 3 (3)
Atrial Arrhythmia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less